CLINICAL TRIAL: NCT00867126
Title: A Pilot Study of Pioglitazone as Second Line Therapy for Patients With Previously Treated Metastatic Adenocarcinoma of the Pancreas With Disease Progression After Gemcitabine Based Chemotherapy
Brief Title: Pioglitazone as Second-Line in Patients With Metastatic Pancreatic Cancer After Treatment With Gemcitabine
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-02208; CDR0000637622 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01036 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: pioglitazone hydrochloride
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Pioglitazone may slow the growth of tumor cells and may be an effective treatment for pancreatic cancer.

PURPOSE: This phase I trial is studying how well pioglitazone works as second-line therapy in treating patients with metastatic pancreatic cancer that progressed after treatment with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To describe changes in markers of insulin resistance, including serum adiponectin levels, standard glucose tolerance testing, and fasting serum glucose and insulin levels, in patients with previously treated metastatic adenocarcinoma of the pancreas treated with pioglitazone hydrochloride as second-line therapy.
* To describe changes in weight in these patients.
* To describe changes in ECOG performance status in these patients.
* To describe changes in symptoms and quality of life of these patients using the validated FACT-Hep scale version 4 questionnaire.

Secondary

* To determine the tumor response as measured by RECIST criteria in these patients.
* To determine the time to disease progression in these patients.

OUTLINE: Patients receive oral pioglitazone hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients complete a quality-of-life questionnaire at baseline, every 4 weeks during therapy, and then at the completion of therapy.

Patients undergo blood sample collection at baseline, every 4 weeks during therapy, and then at the completion of therapy for laboratory biomarker studies. Samples are analyzed for levels of insulin resistance markers (adiponectin, glucose, and insulin).

After completion of study therapy, patients are followed monthly for 6 months and then every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease
  * Previously treated disease
* Disease progression after first-line gemcitabine hydrochloride-based chemotherapy
* Radiologically measurable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Serum creatinine < 1.5 times upper limit of normal (ULN) OR creatinine clearance > 45 mL/min
* Total bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No NYHA class III-IV congestive heart failure
* No unstable angina
* No second malignancy except for localized nonmelanoma skin cancer
* No psychiatric or addictive disorders that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* Prior systemic therapy with fluorouracil, capecitabine, oxaliplatin, or erlotinib hydrochloride allowed
* More than 12 months since prior and no other concurrent thiazolinediones
* More than 6 months since prior treatment with immunosuppressive or immunomodulatory agents
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Insulin resistance markers as measured by standard glucose tolerance testing and serum adiponectin levels at baseline, every 4 weeks during therapy, and then at the completion of therapy
Fasting serum glucose and insulin levels as measured at baseline, every 4 weeks during therapy, and then at the completion of therapy
Changes in weight as measured at baseline, every 4 weeks during therapy, at the completion of therapy, and then monthly for 6 months and every 3 months for 2 years
Changes in ECOG performance status as measured at baseline, weekly during the first course of therapy, every 4 weeks during the rest of therapy, at the completion of therapy, and then monthly for 6 months and every 3 months for 2 years
Changes in symptoms and quality of life as measured by the validated FACT-Hep scale version 4 questionnaire at baseline, every 4 weeks during therapy, and then at the completion of therapy

SECONDARY OUTCOMES:
Objective response (confirmed complete or partial response) as measured by RECIST criteria
Time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Yull E. Arriaga, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States